CLINICAL TRIAL: NCT04554654
Title: The Correlation of Serum Progesterone Levels With the Degree of Endometrial Compaction on the Day of Frozen Embryo Transfer
Brief Title: Progesterone Levels and Endometrial Compaction in Frozen-Thawed Embryo Transfer Cycles
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cem Demirel (Other)
Responsible Party: Sponsor-Investigator, Cem Demirel, professor doctor, Memorial Ataşehir Hospital
Organization: Memorial Ataşehir Hospital (Other)
Other Study IDs: 9995381
Record Dates: First submitted 2020-09-04; First posted 2020-09-18 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Infertility, Female; Infertility of Uterine Origin; Implantation; Placenta
Keywords: frozen-thawed embryo transfer; endometrial compaction; progesterone
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- frozen embryo transfer cycles: patients undergoing frozen embryo transfer with artificial hormone replacement
  Interventions: Diagnostic Test: transvaginal ultrasound,

INTERVENTIONS:
Diagnostic Test: transvaginal ultrasound, — transvaginal ultrasound performed on day of the start of progesterone supplementation and on the day of frozen embryo transfer; serum progesterone level measurement on day of frozen embryo transfer
  Other Names: serum progesterone level measurement

SUMMARY:
This study is intended to determine whether there is a correlation between endometrial compaction and serum progesterone levels on the day of frozen embryo transfers by using transvaginal sonography for the endometrial assessment.

DETAILED DESCRIPTION:
This study is planned to be conducted by prospectively evaluating approximately 200 frozen embryo transfers within 6 months in a single center. Patients planned to be included in the study are started estrodiol 6 mg / day on day2-3 of mensturation. 12 days after the start of estrogen, patients who have endometrial thickness over 7 mm are then started vaginal progesterone supplementation as per routine practice and are eventually proceeded to embryo transfer either on day 4 or 6 of progesterone supplementation. In this study investigators are intended to measure endometrial thickness transvaginally on the day of embryo transfer to accurately determine the presence of endometrial compaction, assess serum progesterone levels, evaluate any possible correlations between endometrial compaction, serum progesterone levels and pregnancy rates.

ELIGIBILITY:
Inclusion Criteria:

1. Woman aged 20-40 years
2. Hormonal(estrogen and progesterone) frozen- thawed embryo transfer cycles
3. Having available blastocyst(s) cryopreserved by vitrification method.

Exclusion Criteria:

1. Recurrent implantation failure
2. Recurrent pregnancy loss
3. Presence of uterine pathology
4. Requirement for fresh embryo(s);
5. Presence of any clinically relevant systemic disease contraindicated for assisted reproduction or pregnancy
6. Allergy history for relevant drugs
7. Body mass index of <18 or >38 kg/m2 at screening
8. Current breastfeeding or pregnancy
9. Refusal or inability to comply with the requirements of the protocol for any reason, including scheduled clinic visits and laboratory tests
10. Natural or modified natural cycles

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female patients underwent infertility treatment
Study Population: Women underwent frozen embryo transfer
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-01-15 (Estimated); Study Completion 2021-02-15 (Estimated)

PRIMARY OUTCOMES:
Ongoing pregnancy rates | 12 weeks after the last menstrual period of the patient
  Presence of at least one live fetus at the end of the 12th gestational week in patients with endometrial compaction compared to patients without endometrial compaction after frozen embryo transfer

SECONDARY OUTCOMES:
The Correlation of Serum Progesterone Levels With the Degree of Endometrial Compaction on the Day of Frozen Embryo Transfer | On the day of frozen embryo transfer
  endometrium compacted (became thinner) after the administration of progesterone
Clinical pregnancy rate | 6-7 weeks after the last menstrual period of the patient
  Presence of an intrauterine gestational sac with fetal heart beat at 7th week of gestation
Implantation rate | 5 weeks after the last menstrual period of the patient
  Percentage of gestational sacs compared to the number of embryos transferred
Clinical miscarriage rate | after 5th gestational week
  pregnancy loss after ultrasonographic detection of an intrauterine gestational sac

CONTACTS AND LOCATIONS:
Locations (1):
- Ataşehir Memorial Hospital IVF Department, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No